CLINICAL TRIAL: NCT01376206
Title: Drug Use Investigation for ALLERMIST
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113407
Record Dates: First submitted 2011-06-09; First posted 2011-06-20 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Rhinitis
MeSH Terms: conditions — Rhinitis | interventions — Fluticasone

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects prescribed ALLERMIST: Subjects with allergic rhinitis prescribed ALLERMIST during study period
  Interventions: Drug: Fluticasone

INTERVENTIONS:
Drug: Fluticasone — Collection of safety data

SUMMARY:
To investigate possible problems or questions in safety and efficacy of ALLERMIST Nasal Spray in Japanese subjects with allergic rhinitis under the practical use conditions

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of allergic rhinitis
* Use ALLERMIST for the first time
* Expected to use ALLERMIST for long-term (1 year)

Exclusion Criteria:

* Subjects with infection which fluticasone is not effective
* Subjects with deep mycosis
* Subjects with hypersensitivity to fluticason

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who have allergic rhinitis for which the indication of ALLERMIST has been approved and who are using ALLERMIST for the first time.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2009-12; Primary Completion 2010-09 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
The number of adverse events in Japanese subjects with allergic rhinitis treated with fluticasone nasal spray | Four weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline